CLINICAL TRIAL: NCT06048536
Title: An Open-label, Phase II, Dose-finding Study of Three Dose Strengths of MR-130A-01 Contraceptive Transdermal Patch in Healthy Pre-menopausal Women
Brief Title: Dose-finding Study of MR-130A-01 Contraceptive Transdermal Patch
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mylan Pharmaceuticals Inc (Industry)
Responsible Party: Sponsor
Organization: Viatris Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MR-130A-01-TD-2001
Record Dates: First submitted 2023-05-08; First posted 2023-09-21 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Contraception

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Norelgestromin low dose 2.43mg 28/0 regimen non-Obese (Experimental)
  Interventions: Drug: MR-130A-01 Transdermal patch
- Norelgestromin mid dose 3.64mg 28/0 regimen non-Obese (Experimental)
  Interventions: Drug: MR-130A-01 Transdermal patch
- Norelgestromin high dose 4.86mg 28/0 regimen non-Obese (Experimental)
  Interventions: Drug: MR-130A-01 Transdermal patch
- Norelgestromin high dose 4.86mg 21/7 regimen non-Obese (Experimental)
  Interventions: Drug: MR-130A-01 Transdermal patch
- Norelgestromin mid dose 3.64mg 28/0 regimen Obese (Experimental)
  Interventions: Drug: MR-130A-01 Transdermal patch
- Norelgestromin high dose 4.86mg 28/0 regimen Obese (Experimental)
  Interventions: Drug: MR-130A-01 Transdermal patch
- Norelgestromin high dose 4.86mg 21/7 regimen Obese (Experimental)
  Interventions: Drug: MR-130A-01 Transdermal patch

INTERVENTIONS:
Drug: MR-130A-01 Transdermal patch — MR-130A-01 transdermal patch, containing 2.43 mg Norelgestromin, will be worn 28 days per cycle with no patch free period.
  Arms: Norelgestromin low dose 2.43mg 28/0 regimen non-Obese
Drug: MR-130A-01 Transdermal patch — MR-130A-01 transdermal patch, containing 3.64 mg Norelgestromin, will be worn 28 days per cycle with no patch free period.
  Arms: Norelgestromin mid dose 3.64mg 28/0 regimen Obese; Norelgestromin mid dose 3.64mg 28/0 regimen non-Obese
Drug: MR-130A-01 Transdermal patch — MR-130A-01 transdermal patch containing 4.86 mg Norelgestromin, will be worn 28 days per cycle with no patch free period
  Arms: Norelgestromin high dose 4.86mg 28/0 regimen Obese; Norelgestromin high dose 4.86mg 28/0 regimen non-Obese
Drug: MR-130A-01 Transdermal patch — MR-130A-01 Transdermal patch MR-130A-01 transdermal patch containing 4.86 mg Norelgestromin, will be worn 21 days with a 7-day patch free period.
  Arms: Norelgestromin high dose 4.86mg 21/7 regimen Obese; Norelgestromin high dose 4.86mg 21/7 regimen non-Obese

SUMMARY:
A single-center, randomized, open-label, parallel-group, multi-arm, phase II clinical trial in healthy women aged 18 to 35 years who have a documented ovulatory cycle prior to randomization.

DETAILED DESCRIPTION:
MR-130A-01 is a progestin-only TDS containing NGMN as its progestin. NGMN is currently available in combination with EE in CHC TDSs Xulane® (US) and Evra® (EU), at doses of 150 mcg/day (Xulane® USPI 2022) and 203 mcg/day (Evra®SmPC 2022) respectively. In the currently planned dose-finding clinical trial the ovulation inhibition and the impact on further physiological functions and hormones of the three dose strengths of MR-130A-01 will be investigated in healthy pre-menopausal obese and non-obese women with ovulatory menstrual cycles. Eligible subjects will be randomized according to their body mass index (BMI) into one of 7 treatment arms with different doses and regimens of IMP administration. The IMPs which are transdermal patches, will be applied to the skin (upper outer arm, abdomen, buttock or back) and will be changed weekly. Depending on the treatment arm, either 4 or 3 patches of an allocated patch strength will be applied per cycle (28/0-day regimen and 21/7-day regimen). Patch adhesion will be assessed by the subjects daily and the results (adhesion scores) will be recorded in a diary. Throughout the clinical trial, ovarian activity will be monitored by TVUS, and blood samples will be collected for determination of progesterone (P), estradiol (E2), LH and FSH concentrations. The inhibition of ovulation will be assessed by Hoogland and Skouby Score (HSS). In addition, bleeding pattern will be assessed based on the subject's records of bleeding and its intensity in a diary.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy, post-menarcheal and premenopausal women of age 18 to 35 years inclusive).
2. BMI ≥18.0 kg/m2 at screening examination.
3. Subjects must be in good physical and mental health as determined by vital signs, medical history, and physical and gynecological examination, as assessed by the investigator.
4. Written informed consent, after having been informed about benefits and potential risks of the clinical trial, as well as details of the insurance taken out to cover the subject participating in the clinical trial.
5. Status at least 3 months after a delivery, abortion, and stopping lactation, if applicable, before screening.
6. Has regular menstrual cycles that are between 21 and 35 days in duration as reported by the subject during anamnesis, with an intact uterus and ovaries. If the subject uses hormonal birth control at screening, historic data should be used to evaluate this criterion.
7. Both ovaries must be visible on TVUS examination during screening.
8. Ovulatory pre-treatment cycle, as confirmed by a progesterone concentration >10.0 nmol/L.
9. Subjects must consent to use reliable non-hormonal contraceptive methods (male condoms, diaphragm, or heterosexual abstinence) throughout the study, unless the subject has a history of female sterilization or sterilization of the sexual partner.

Exclusion Criteria:

1. Known hypersensitivity or intolerance to any ingredient of the investigational product.
2. History or presence of dermal sensitivity to medicated patches or to topical applications including bandages, surgical tape.
3. Pregnancy or a positive serum beta human chorionic gonadotropin (β-hCG) pregnancy test at screening.
4. Clinically relevant abnormal findings from serum biochemistry and hematology and HBsAg and Hepatitis C virus/human immunodeficiency virus (HIV) serology as evaluated by the investigator.
5. ASAT (aspartate-aminotransferase) > 20 % upper limit of normal (ULN), ALAT (alanine-aminotransferase) > 10 % ULN, bilirubin > 20% ULN (except in case of existing Morbus Gilbert-Meulengracht deduced from anamnesis/medical history) and creatinine > 0.1 mg/dL ULN (limit of > 0.1 mg/dL corresponds to > 9 μmol/l ULN).
6. Use of a non-hormonal intra-uterine device within the pre-treatment cycle or any hormonal contraception as follows:

   * Short-acting hormonal contraceptives such as oral, patch, ring or intra-uterine systems within the menstrual cycle prior to the pre-treatment cycle.
   * Injectable (intramuscularly or subcutaneously) within 10 months (three-month treatment duration), 6 months (two-month treatment duration) or 3 months (one-month treatment duration) prior to the start of pre-treatment cycle or implants within the menstrual cycle prior to the pre-treatment cycle.
7. Known or suspected malignancy or history thereof.
8. Has unexplained vaginal bleeding within the past 6 months suspicious for serious condition, or any abnormal bleeding which is expected to recur during the study (eg. bleeding from cervical polyp, recurrent bleeding after sex).
9. History or presence of ischemic heart disease, coronary artery disease, myocardial infarction, stroke, other cerebrovascular diseases including transient ischemic attacks (TIAs).
10. Known dyslipidemias with other known cardiovascular risk factors.
11. History or presence of hypertension (including adequately controlled hypertension) or hypertension with vascular disease or elevated blood pressure (BP) defined as systolic BP ≥140 mm Hg or diastolic BP ≥90 mm Hg, measured in sitting position after at least 5 minutes of rest (a single reading of blood pressure level is not sufficient to classify a woman as hypertensive).
12. Pulse rate < 50 bpm or > 90 bpm
13. Presence of deep vein thrombosis/pulmonary embolism.
14. Has any comorbid condition that may require major surgery with prolonged immobilization during the study period.
15. History or presence of migraine with aura.
16. Presence of liver disease including severe (decompensated) cirrhosis, benign (e.g., hepatocellular adenoma) or malignant liver tumors.
17. Chronic disease potentially necessitating organ transplantation during the anticipated course of the study.
18. Subjects having any other known contraindication to progestin only contraception as defined by category 3 or 4 conditions per World Health Organization Medical eligibility

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 168 (Actual)
Dates: Start 2023-12-22 (Actual); Primary Completion 2024-01-18 (Actual); Study Completion 2024-01-18 (Actual)

PRIMARY OUTCOMES:
Proportion of responder overall (subjects with no ovulation in both treatment cycles) | 56 days
  A responder is a subject with no ovulation. A responder is a subject with no ovulation. Ovulation during treatment is defined as a Hoogland-Skouby score 5 or 6 in combination with fulfilment of Landgren criterion.
Proportion of responder in cycle (subjects with no ovulation in one of the treatment cycles) | 56 days
  A responder is a subject with no ovulation. A responder is a subject with no ovulation. Ovulation during treatment is defined as a Hoogland-Skouby score 5 or 6 in combination with fulfilment of Landgren criterion.

SECONDARY OUTCOMES:
For assessment of ovarian activity, Hoogland and Skouby score frequency analysis will be provided for: | 56 days
  * Subjects with either HSS 5 or 6
  * Subjects with HSS <5
  * Subjects for each HSS from 1 to 6
  * Subjects with HSS 5 or 6 and positive Landgren criterion
  * Subjects with HSS 5 or 6 and negative Landgren criterion.
  Frequency analysis will be provided per treatment arm for each of the treatment cycles.
Corpus luteum function will be evaluated in subjects by using Landgren criteria in conjunction with Hoogland and Skouby score. Frequency analysis will be provided for: | 56 days
  * Subjects with HSS 5 or 6 and positive Landgren criterion
  * Subjects with HSS 5 or 6 and negative Landgren criterion. Frequency analysis will be provided per treatment arm for each of the treatment cycles. Furthermore, frequency of occurrence of any Landgren criterion over both cycles will be calculated.
The diameter of the largest FLS in both the right and left ovary will be measured (for each, the mean diameter from two directions). The largest of all follicles is considered the dominant FLS (FLSdom) for that study day. | 56 days
  From this, the subject-wise maximum FLS diameter (MFD) will be calculated separately for each treatment cycle and over both cycles. The maximum endometrial thickness (ETmax) subject-wise will be calculated for each treatment cycle and for the entire treatment period using transvaginal ultrasound. This will be reported per visit and for each of the treatment cycles
The effect of cervical mucus will be calculated by Insler score. The subject-wise maximum Insler score (ISmax) will be calculated for each treatment cycle and for the entire treatment period. | 56 days
To assess the effects of MR-130A-01 on sexual hormones(estradiol [E2], progesterone [P]) hormone concentrations determined in serum | 56 days
  Descriptive statistics will be given per treatment arm for:
  Concentrations of FSH, LH, E2, and P at each visit
  • Max FSH, max LH, max E2, mean E2, max P in each treatment cycle and over both cycles
Steady state concentration of NGMN and norgestrel will be calculated per treatment arm by means of non-compartmental analysis. | 56 days
  Descriptive statistics (N, arithmetic means, SD, medians, minimum, maximum geometric means, geometric CV) will be presented for all pharmacokinetic parameters, separately for each treatment and analyte.
Patch adhesion will be evaluated by both data subject diary and site personnel. | 56 days
  Frequency analysis of patch adhesion scores will be provided per treatment arm
  * For each day of the application period of one patch (Day 1 to Day 7)
  * For the subject-wise mean and maximum application score over the entire application period of one patch (1 week).
  In addition, the following evaluations will be presented per treatment arm for each evaluation time-point (day/week):
  * Proportion of subjects achieving greater than 90% adherence (score 0)
  * Proportion of subjects with a meaningful degree of detachment (patch detachment ≥25% (estimated score ≥2)
  * Number of patches that are completely detached (score 4).
Safety will be evaluated by TEAEs considering action taken, frequency, seriousness, intensity, relationship to the IMP, outcome as well as treatment. | 56 days
  Evaluation will be described by absolute and relative frequency. Tolerability will be evaluated by application site reactions. Frequency analysis of skin irritation categories will be provided per treatment arm over the entire treatment period.
Bleeding pattern will be assessed in each single subject over treatment cycle 1 and treatment cycle 2 (defined as 56-day reference period) by | 56 days
  * Incidences (percentage of subjects) of unscheduled/scheduled bleeding and/or spotting episodes within the reference period
  * The mean, median and range of number of observed days of bleeding and/or spotting within the reference period
  * The observed days of bleeding and/or spotting within the reference period presented as total days, unscheduled days and scheduled days for bleeding and/or spotting, bleeding only and spotting only
  * Incidences (percentage of subjects) of complete absence of bleeding or spotting during the reference period.

CONTACTS AND LOCATIONS:
Overall Officials: Sandeep Jagtap, Study Director — Mylan Pharmaceuticals Private Limited (A Viatris Company)
Locations (1):
- dinox GmbH, Berlin, Germany